CLINICAL TRIAL: NCT01351727
Title: Epidemiologic Follow Up Study of Newly Diagnosed Epilepsy Among Seniors From Different Ethnic Groups
Brief Title: Epidemiologic Follow Up Study of Newly Diagnosed Epilepsy Among Seniors
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jenny Chong, Research Associate Professor, University of Arizona
Other Study IDs: 10-0916-01
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Epileptic Seizures
Keywords: seniors; seizures; epilepsy; quality of life
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Seniors with Seizures: Seniors aged 65 or older with newly diagnosed seizures (consistent with epilepsy) or epilepsy as of October, 2010.

SUMMARY:
The purpose of this proposed research is to identify individuals in southeastern Arizona aged 65 years and older who have new onset seizures (or newly diagnosed epilepsy) and monitor them for at least two years. In doing so the investigators will be able to describe the public health burden of this condition and to identify factors that predict clinical outcomes and health care needs in this population, using quantitative, administrative, and qualitative data. The aims of this proposed research are 1) to determine the two-year incidence of newly diagnosed epilepsy in the target population, 2) describe health care resource utilization of the target population using Medicare data, 3) validate the use of Medicare beneficiary data to estimate incidence of epilepsy, and 4) describe the burden of this condition in different ethnic groups.

DETAILED DESCRIPTION:
Seniors who have had new onset seizures or newly diagnosed epilepsy will be recruited from emergency departments (EDs), neurology clinics, primary care clinics (including geriatric clinics), and other service providers from networks maintained by the Area Agencies on Aging that serve seniors in southeastern Arizona. Data will be collected in the form of bi-annual surveys,administrative data (from Medicare), in-depth interviews, and focus groups. Medicare data will be used to describe and evaluate the likelihood of being hospitalized or admitted to a long-term facility within two years of being diagnosed, medication adherence and persistence, and comparing the cost of care between the newly-diagnosed seniors with epilepsy and comparable seniors who do not have epilepsy. The feasibility and validity of using the Medicare claims data to estimate newly diagnosed epilepsy will also be assessed. Finally, the impact of epilepsy on health related quality of life, mental health, perceived stigma, and family and caregivers will also be evaluated through surveys and qualitative data collection methods, and ethnic differences will also be described.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* New onset seizure or newly diagnosed epilepsy as of October 2010
* Is a resident of Pima, Cochise or Santa Cruz County

Exclusion Criteria:

* Seizure dues to hyponatremia, hypoglycemia, alcohol use (with no evidence of other seizures)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitals (including emergency departments), neurology specialist clinics, primary care clinics, communities (in Cochise, Pima, Santa Cruz Counties)including nursing homes, skilled nursing facilities, assisted living facilities.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
A two-year incidence rate of new-onset seizures and/or newly-diagnosed epilepsy among seniors in southeastern Arizona. | Up to four years
  A surveillance mechanism will be developed to identify and recruit seniors from emergency departments, neurology clinics, primary care clinics, and other service providers for seniors.

SECONDARY OUTCOMES:
Compare the impact of epilepsy on the different ethnic groups of seniors with epilepsy | Up to four years
  1. Assess the level and ethnic differences in health-related quality of life, mental health, and perceived stigma among seniors with seizures.
  2. Use in-depth interviews to explore issues related to epilepsy and its treatment.
  3. Conduct focus groups with caregivers to learn about their concerns and barriers.

CONTACTS AND LOCATIONS:
Overall Officials: David Labiner, MD, Principal Investigator — University of Arizona; Jenny Chong, PhD, Principal Investigator — University of Arizona
Locations (1):
- Pima, Cochise, Santa Cruz Counties, Tucson, Arizona, United States

REFERENCES:
- [Background] Martin R, Vogtle L, Gilliam F, Faught E. What are the concerns of older adults living with epilepsy? Epilepsy Behav. 2005 Sep;7(2):297-300. doi: 10.1016/j.yebeh.2005.05.003. PMID 15996527
- [Background] Pallin DJ, Goldstein JN, Moussally JS, Pelletier AJ, Green AR, Camargo CA Jr. Seizure visits in US emergency departments: epidemiology and potential disparities in care. Int J Emerg Med. 2008 Jun;1(2):97-105. doi: 10.1007/s12245-008-0024-4. Epub 2008 Jun 5. PMID 19384659
- [Background] Tallis R, Hall G, Craig I, Dean A. How common are epileptic seizures in old age? Age Ageing. 1991 Nov;20(6):442-8. doi: 10.1093/ageing/20.6.442. PMID 1776595